CLINICAL TRIAL: NCT03919396
Title: Effectiveness of Myopia Control by Breath-O Correct Orthokeratology Lenses in Different Myopia Progression Groups
Brief Title: Effectiveness of Myopia Control by Breath-O Correct Orthokeratology Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: SEED Co. Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HongKongPU_Optometry3
Record Dates: First submitted 2019-04-16; First posted 2019-04-18 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2021-08

CONDITIONS: Myopia; Orthokeratology
Keywords: Myopia; Myopia Control; Orthokeratology; Electroretinogram; Multifocal Electroretinogram
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OrthoK (orthokeratology) (Experimental): Group wearing Breath-O corrected orthokeratology lenses for 2 years
  Interventions: Device: Breath-O orthokeratology lenses
- SV Lenses (Single vision) (No Intervention): Group wearing spectacle with single vision lenses for 2 years

INTERVENTIONS:
Device: Breath-O orthokeratology lenses — Specially designed rigid gas permeable lenses which
  1. reshapes corneal profile for myopia control
  2. has higher elasticity compared to traditional lens material.
  Arms: OrthoK (orthokeratology)

SUMMARY:
This is a 24-month longitudinal randomized controlled trial aiming to evaluate the effectiveness of myopia control by Breath-O correct orthokeratology lenses in different myopia progression groups classified according to their initial electro-retinal responses.

DETAILED DESCRIPTION:
Myopia is the most common refractive error in the world. In Hong Kong, the number of children in myopia is on the rise and approximately 80% of children are myopic by the end of childhood. Orthokeratology is one of the most successful myopia control methods adopting the strategy of peripheral defocus, in which the natural emmetropization process is harnessed by the myopic defocus induced by the orthokeratology lenses.Currently, Breath-O correct lenses are new designed ready-made orthokeratology lenses which are made of new material with higher elasticity as compared traditional lens material.

A recent study has shown young children with an initial weakened central electrical signal from the inner retina had faster myopia progression as measured by multifocal electroretinogram(ERG). We will classify the slow and fast progression group based on the ERG results, so as to evaluate the clinical effectiveness of the newly designed lenses in controlling myopia in children with different rates of progression.

ELIGIBILITY:
Inclusion Criteria:

* Refractive error: Spherical: -1.00D to -4.00D; Cylindrical: half of Sph (against-the-rule Astig.: less than -0.75D)
* Best corrected Visual acuity: monocular ETDRS 0.1 or better

Exclusion Criteria:

* Ocular abnormality
* Contra-indicated for overnight orthokeratology lens wear
* History of refractive surgery
* Systemic diseases
* History of orthokeratology lenses wearing or other myopia control methods

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Subjective Refraction | up to 24 months
  Refractive Error ( in Diopter )

SECONDARY OUTCOMES:
Axial Length | up to 24 months
  Length of eye ball

CONTACTS AND LOCATIONS:
Overall Officials: Henry HL Chan, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- School of Optometry, Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No